CLINICAL TRIAL: NCT05186324
Title: Fabry Patient's Experience Of PegunigaLsidasE Alfa Monthly Infusion - PEOPLE Study
Brief Title: Fabry Patient's Experience Of PegunigaLsidasE Alfa Monthly Infusion
Acronym: PEOPLE
Status: Completed | Type: Observational
Sponsor: Chiesi Farmaceutici S.p.A. (Industry)
Collaborators: Protalix (Industry); Iqvia Pty Ltd (Industry)
Responsible Party: Sponsor
Other Study IDs: CLI-06657AA1-05
Record Dates: First submitted 2021-12-21; First posted 2022-01-11 (Actual); Last update posted 2023-03-21 (Actual); Status verified 2023-03

CONDITIONS: Fabry Disease
MeSH Terms: conditions — Fabry Disease | interventions — Interviews as Topic

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Interview — During each interview, patients will be asked questions to collect demographic and clinical information, and asked a set of open-ended questions with probes to describe their experiences with Fabry disease (symptomology and impacts on patient's lives [i.e., activities of daily living, school/work, ability to take holidays/vacation]), and pegunigalsidase alfa treatment (experience of infusions and schedule) and their experience of change in symptoms and impacts over the BRIGHT-F51 clinical study.
  A semi-structured discussion guide will be used to conduct the approximately 60-minute interviews. The use of open-ended questions avoids bias and questions will not be read verbatim to allow for a free-flowing discussion.

SUMMARY:
Pegunigalsidase alfa (PRX-102) is a long-term enzyme replacement therapy design for the treatment of patients with Fabry disease. Although in the clinical development program patient-reported outcomes and clinician-reported outcomes have been included, this may not allow for a sufficiently accurate assessment of the quality of life in patients with Fabry Disease treated with pegunigalsidase alfa.

This study will collect the patient experience on the pegunigalsidase alfa treatment administered intravenously every 4 weeks in the BRIGHT-F51 clinical study (NCT03614234).

DETAILED DESCRIPTION:
This is an additional qualitative concept elicitation interview-based study to further understand the patients' experience with Fabry disease and with the pegunigalsidase alfa administered intravenously every 4 weeks. Patients will be asked a set of open-ended questions with probes to describe their experiences with Fabry disease on treatment with pegunigalsidase alfa. Qualitative research methods will be used to obtain a deeper understanding of the patient experience by generating in-depth information about the experiences, perspectives, and feelings of patients and others, in their own words (FDA Patient-Focused Drug Development Guidance 2).

The study will be offered to the 29 patients participating in the BRIGHT-F51 clinical trial (NCT03614234).

ELIGIBILITY:
Inclusion Criteria:

* The patient is participating in study PB-102-F51
* The patient is willing and able to participate in a 60-minute recorded interview
* The patient is able to read, understand, and speak sufficiently to participate in the interviews
* The patient signs informed consent to participate in the study

Exclusion Criteria:

* At investigators discretion, patient is considered to be unable to participate in a 60- minute telephone interview.
* Patient has any clinically relevant medical or psychiatric condition that, in the opinion of the investigator would interfere with the completion of the study activities. This includes but is not limited to language, speech, hearing or cognitive disorders that could impact a patient's ability to participate in an interview-based discussion.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The PEOPLE study will recruit patients who have taken part in the BRIGHT (F50) clinical trial and are participating in the BRIGHT-F51 extension clinical trial (regardless of their infusion schedule and dosing regimen). Based on the total number of patients (n=29) enrolled in the BRIGHT-F51 clinical trial extension, up to 29 patients could be recruited.
Sampling Method: Non-Probability Sample
Enrollment: 23 (Actual)
Dates: Start 2022-01-26 (Actual); Primary Completion 2022-08-31 (Actual); Study Completion 2022-08-31 (Actual)

PRIMARY OUTCOMES:
Symptoms experience while on treatment with pegunigalsidase alfa | 2 years
  Description of the symptoms experienced by patients treated with pegunigalsidase alfa for more than 2 years
Change in symptoms experienced | 2 years
  Description of any worsening or relapse in Fabry disease symptoms during the 4 weeks between two consecutive infusions of pegunigalsidase alfa administered every 4 weeks in patients treated for more than 2 years
Impacts of Fabry disease on patient's life | 2 years
  Description of the impacts of Fabry disease on patient's lives i.e., activities of daily living, school/work, ability to take holidays/vacation) in patients treated with pegunigalsidase alfa for more than 2 years
Change in the ability to perform daily activities | 2 years
  Description of any worsening or relapse in the ability to perform daily activities during the 4 weeks between two consecutive infusions of pegunigalsidase alfa in patients treated every 4 weeks for more than 2 years
Patients' perceptions of the advantages and disadvantages associated with the every 4 weeks infusion schedule | 2 years
  Summary of patients' perceptions of the advantages and disadvantages associated with the every 4 weeks infusion schedule (compared to the 2-week infusion schedule) in patients treated with pegunigalsidase alfa for more than 2 years

OTHER OUTCOMES:
Perception of change in symptoms and impacts with infusion schedules | 2 years
  Description of patients' perception of change in symptoms and impacts with the with the every 4 weeks infusion schedule compared to the 2-week infusion schedule in patients treated with pegunigalsidase alfa for more than 2 years

CONTACTS AND LOCATIONS:
Locations (12):
- United States (7):
  - #02, Birmingham, Alabama
  - #03, Atlanta, Georgia
  - #04, Iowa City, Iowa
  - #11, Grand Rapids, Michigan
  - #06, Dallas, Texas
  - #05, Salt Lake City, Utah
  - #01, Fairfax, Virginia
- #22, Antwerp, Belgium
- #50, Copenhagen, Denmark
- #56, Napoli, Italy
- United Kingdom (2):
  - #28, Cambridge
  - #07, London

IPD SHARING:
Plan to Share IPD: No